CLINICAL TRIAL: NCT06979206
Title: Effects of Binaural Beats on Inhaled Anesthetic Requirements During General Anesthesia in Pediatric Patients: A Prospective, Randomized Controlled Trial
Brief Title: Effects of Binaural Beats on Inhaled Anesthetic Requirements During General Anesthesia in Pediatric Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ji-Hyun Lee, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2501-127-1610
Record Dates: First submitted 2025-05-11; First posted 2025-05-18 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: General Anesthesia; Children

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Binarual beat group (Experimental): In this group, a binaural beat audio file is applied throughout the maintenance of anesthesia. The binaural beat consists of pure tones at 431 Hz in the left ear and 432 Hz in the right ear, delivered via earphones continuously until the end of anesthesia. Anesthesia is maintained with sevoflurane, and its concentration is adjusted to maintain a Patient State Index (PSI; SEDLine®; Masimo Corp., Irvine, USA) between 20 and 50. At the end of surgery, sevoflurane administration is discontinued, and ondansetron 0.1 mg/kg, acetaminophen 15 mg/kg, ketorolac 0.5 mg/kg, and a neuromuscular reversal agent are administered to facilitate emergence from anesthesia.
  Interventions: Other: Application of Binarual Beat
- Control group (No Intervention): This group undergoes anesthesia using the conventional method, with maintenance of anesthesia achieved using sevoflurane. The concentration of sevoflurane is adjusted to maintain a Patient State Index (PSI; SEDLine®; Masimo Corp., Irvine, USA) between 20 and 50. At the end of surgery, sevoflurane administration is discontinued, and ondansetron 0.1 mg/kg, acetaminophen 15 mg/kg, ketorolac 0.5 mg/kg, and a neuromuscular reversal agent are administered to facilitate emergence from anesthesia.

INTERVENTIONS:
Other: Application of Binarual Beat — The binaural beat audio file consists of pure tones at 431 Hz in the left ear and 432 Hz in the right ear, delivered via earphones continuously until the end of anesthesia.
  Arms: Binarual beat group

SUMMARY:
The hypothesis of this study is that continuously delivering binaural beats with a phase difference corresponding to the slow-delta frequency band during anesthesia in pediatric patients can clinically and significantly reduce the required dose of the commonly used inhalational anesthetic, sevoflurane. To test this hypothesis, the study will compare the average end-tidal concentration of sevoflurane between a group exposed to continuous binaural beats (approximately 1 Hz phase difference) during surgery and a control group not exposed to such auditory stimulation.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients under 3 years of age undergoing superficial surgery lasting more than 1 hour under general anesthesia (e.g., nevus excision, polydactyly/syndactyly surgery, dermoid cyst excision, thyroglossal duct cyst excision, preauricular fistula excision, inguinal hernia repair, orchiopexy, other mass excisions, strabismus surgery, etc.).
2. American Society of Anesthesiologists (ASA) physical status classification I or II.

Exclusion Criteria:

* Neonates or premature infants
* Children with hearing impairment or currently using hearing aids
* Children with neurological disorders
* Children with respiratory diseases
* Children undergoing neurosurgery or cardiac surgery
* Other patients deemed inappropriate for inclusion in the clinical trial at the discretion of the investigator or study staff

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2025-05-30 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
The average EtSevo (end-tidal sevoflurane concentration, vol%) maintained during surgery. | During surgery, more than 1 hour